CLINICAL TRIAL: NCT02632695
Title: Physical Activity Interventions for Leg Ulcer Patients
Acronym: FOOTFIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Teresa Kelechi, Professor, Medical University of South Carolina
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00043451
Record Dates: First submitted 2015-12-01; First posted 2015-12-17 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-05

CONDITIONS: Leg Ulcers; Venous Ulcers; Varicose Ulcers
MeSH Terms: conditions — Leg Ulcer; Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FOOTFIT Plus (Experimental): The intervention consists of: 1) a prescribed, evidence-based, phased, non-exertive physical activity conditioning activities for lower leg function (CALF) movements that are to be performed daily at home; 2) a low-cost, tri-axial Bluetooth® enabled highly sensitive motion-sensing accelerometer and tracking device (BEAT) worn on the foot during CALF to capture frequency and intensity of foot movements; and 3) a Smartphone that receives foot movement data, provides automated educational/motivational messages, and reports and allows regular communication with the wound care provider on progress.
  Interventions: Device: FOOTFIT
- FOOTFIT (Experimental): The intervention consists of: 1) a prescribed, evidence-based, phased, non-exertive physical activity conditioning activities for lower leg function (CALF) movements that are to be performed daily at home; 2) a low-cost, tri-axial Bluetooth® enabled highly sensitive motion-sensing accelerometer and tracking device (BEAT) worn on the foot during CALF to capture frequency and intensity of foot movements; and 3) a Smartphone that receives foot movement data, provides automated educational/motivational messages, and reports. There is not regular communication with the wound care provider on progress.
  Interventions: Device: FOOTFIT

INTERVENTIONS:
Device: FOOTFIT — Individuals with venous leg ulcers will be instructed on physical activity movements for their lower legs to be performed over six weeks while wearing a foot based activity monitor (accelerometer) that will send them motivational messages and progress reports. For those in the FOOTFIT Plus group, individuals will have the option to communicate with their wound care provider via text messages, emails or phone calls.

SUMMARY:
The goal of this study is to test FOOTFIT and enhanced FOOTFIT+, home-based mobile health (mHealth) physical activity (PA) interventions for a minimally ambulatory, chronically-ill, population with leg ulcers. A highly sensitive clinically designed Bluetooth® enabled accelerometer and tracking device (BEAT) worn on the foot during a progressive and evidence-based non-exertive leg conditioning activities for lower leg function (CALF) captures minute foot movements and sends the data to a Smartphone. This six-week feasibility study will compare FOOTFIT to FOOTFIT+, with the added connectivity feature, to promote patient-provider communication, evaluate adherence to PA, and assess signals of efficacy on functional outcomes in a very low fitness population.

DETAILED DESCRIPTION:
FOOTFIT is a study of a lower leg conditioning mHealth intervention for patients with venous leg ulcers. The aims are to compare two versions, one of which is enhanced (FOOTFIT+), to determine which has the greatest impact on physical activity adherence, patient-provider communication, and leg function. FOOTFIT and FOOTFIT+ share three components: 1) a low-cost, tri-axial Bluetooth® enabled highly sensitive accelerometer and tracking device (BEAT) worn on the foot during, 2) phased conditioning activities for lower leg function (CALF) tracked by a, 3) Smartphone that captures signals from BEAT, provides motivational messages, CALF instruction, and automated feedback on progress. Forty patients will be targeted in this six-week study, 20 of which will receive FOOTFIT and 20 FOOTFIT+.

ELIGIBILITY:
Inclusion Criteria:

* Active venous leg ulcer
* Ankle brachial index 0.80 to 1.3 mmHg, a measure of arterial sufficiency
* Sedentary-able to only walk a few steps at a time or not farther than 10 feet
* Not currently exercising or participate in a PA or physical therapy program
* Receives at least weekly wound care anticipated to last for at least six weeks from start of study
* Able to don accelerometer - if unable to apply independently, has assistance from other
* Capable of using Smartphone

Exclusion Criteria:

* Co-morbid conditions such as stroke (limits ankle function)
* Ulcer from other causes (arterial, diabetic, trauma, surgery)
* Documented cognitive impairment (MiniCog)
* No 3G service in area where patient resides

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-04; Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
FOOTFIT feasibility | 6 weeks
  Measure adherence by recording frequency and intensity of foot/toe movements reported in minutes.
FOOTFIT reach | 6 weeks
  Measure reach, recorded as qualitative documents on a log of how patients learned about the study.
FOOTFIT technology implementation procedures | 6 weeks
  Record on study log the number and types of problems encountered with the study nurses teaching participants to use the foot accelerometer technology, the number and types problems reported by patient, the number and types of recommendations made by the participant regarding the use of the accelerometer, and nurse or provider recommendations for changes to refine the foot accelerometer technology, and the number and types of refinements to the technology that were made.
FOOTFIT acceptability | 6 weeks
  Record on study logs the the number (frequency) and types of interactions such as phone calls, emails or texts, between the patient and provider regarding FOOTFIT+ including reasons (i.e., exercises, adverse events that are related to, and not related to the use of the accelerometer).

SECONDARY OUTCOMES:
Efficacy on pain | 6 weeks
  Obtain estimates of variability for short-term functional impacts on pain using the numerical rating scale (NRS) as a single score.
Efficacy on foot strength | 6 weeks
  Obtain estimates of variability for short-term functional impacts on foot strength using the dynamometer and reported as pounds per square inch.
Efficacy on foot range of motion. | 6 weeks
  Obtain estimates of variability for short-term functional impacts on foot range of motion using the goniometer and reported in degrees.
Efficacy on walking function. | 6 weeks
  Obtain estimates of variability for short-term functional impacts on walking function using the Foot and Ankle Ability Measure and reported as a sum score.
Efficacy on walking performance | 6 weeks
  The Six Minute Walk Test reported as distance in feet over six minutes time.

CONTACTS AND LOCATIONS:
Overall Officials: Moby Madisetti, MS, Study Director — Medical University of South Carolina
Locations (1):
- Spartanburg Regional Medical Center, Spartanburg, South Carolina, United States

REFERENCES:
- [Derived] Kelechi TJ, Prentice MA, Mueller M, Madisetti M, Vertegel A. A Lower Leg Physical Activity Intervention for Individuals With Chronic Venous Leg Ulcers: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2020 May 15;8(5):e15015. doi: 10.2196/15015. PMID 32412419